CLINICAL TRIAL: NCT01760616
Title: A Prospective, Multicenter, Open-labeled, Parallel -Controlled Clinical Study Investigating Huaier Granule for Prevention of Disease Progression of Hepatocarcinoma After Non-radical Hepatectomy
Brief Title: Huaier Granule for Prevention of Disease Progression of Hepatocarcinoma After Non-radical Hepatectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficult to recruit patients
Sponsor: Qidong Gaitianli Medicines Co., Ltd (Industry)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-201102
Record Dates: First submitted 2013-01-01; First posted 2013-01-04 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Hepatic Carcinoma
Keywords: Huaier Granule;; After non-radical hepatectomy;; Prevention of Disease Progression of Hepatocarcinoma;; Safety.
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental): Test group: Adjuvant therapy + Huaier Granule group.Administration: the Huaier Granule Electuary should be orally taken from the 15th day after surgery. Usage: Huaier Granule Electuary is continuously taken three times per day, 20g per time, until 144 weeks after surgery or until study termination Adjuvant therapy: the adjuvant therapies are not limited, and for example, all the following treatments can be applied according to the individual's condition and guidelines of the research center: ablation therapy, immunotherapy, chemotherapy, radiotherapy, and Chinese herbs, as well as programs and medications that are used for post-operative liver protection and antiviral treatment
  Interventions: Drug: Huaier Granule
- Control group: adjuvant therapy (No Intervention): Control group: adjuvant therapy Adjuvant therapy: the adjuvant therapies are not limited, and for example, all the following treatments can be applied according to the individual's condition and guidelines of the research center: ablation therapy, immunotherapy, chemotherapy, radiotherapy, and Chinese herbs, as well as programs and medications that are used for post-operative liver protection and antiviral treatment.

INTERVENTIONS:
Drug: Huaier Granule — Huaier Granule is a Chinese medicine, specifications: 20g / bag, manufacturer: Qidong Gaitianli Medicines Co., Ltd..
  Arms: Test group

SUMMARY:
To evaluate the efficacy and safety of Huaier Granule for prevention of disease progression of hepatocarcinoma after non-radical hepatectomy.

DETAILED DESCRIPTION:
A Prospective, Multicenter, Open-labeled, Parallel -controlled Clinical Study, to evaluate the efficacy and safety of Huaier Granule for prevention of disease progression of hepatocarcinoma after non-radical hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 and ≤ 75 years, both male and female;
2. Non-radical hepatectomy has been performed for hepatocellular carcinoma;
3. The hepatocellular carcinoma has been confirmed by pathological examination;
4. The liver and kidney function satisfies the following conditions within 15 days after surgery (excluding day 15): aspartate aminotransferase(AST), glutamic-oxalacetic transaminase(ALT)<3 upper limit of normal(ULN), total bilirubin ≤2 ULN, serum creatinine <1.5 ULN;
5. Other laboratory tests meet the following requirements within 15 days after surgery (excluding day 15): Hb≥9g/dl, platelet count≥60×109/L, neutrophil count> 1.5×109/L;
6. The expected survival time ≥12 weeks;
7. The subjects volunteer to sign the informed consent.

Exclusion Criteria:

1. Non-hepatocellular carcinoma patients;
2. Those who received radical hepatectomy;
3. Those with hepatic decompensation;
4. Pregnant or lactating women;
5. Those with HIV infection or AIDS-associated diseases;
6. Those with severe acute and chronic diseases, such as infection, diabetes cardiac insufficiency, pulmonary insufficiency, renal insufficiency;
7. Those who can not take drugs by oral route; or those develop serious adverse drug reaction;
8. Drug abusers or those with psychological or mental diseases that may interfere with study compliance;
9. Conditions that are considered not suitable for this study investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2015-08-15 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Time to significant progression after surgery and postoperative survival period. | 3 years
  Time to significant progression after surgery, including recurrence of local tumor, intrahepatic and extrahepatic metastasis, etc; and to evaluation of postoperative survival period.

SECONDARY OUTCOMES:
ECOG and QLQ-C30 scores | Week 8, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144
  On week 8, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132 and 144, assess the scores of Eastern Cooperative Oncology Group(ECOG) and quality of life questionnaire(QLQ)-C30 scale.
Iconography assessment | Week 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144
  On week 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132 and 144, give examination of B ultrasonic for Liver, X-ray for chest. If there is a suspected recurrence or metastases, will give enhancement CT/MRI examination for liver and chest; if no recurrence or metastases, will at least give enhancement CT/MRI examination for liver and chest every year.
Alpha-fetoprotein quantitation and related biochemical indicators | Week 8, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144
  On week 8, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132 and 144, monitor Alpha-fetoprotein quantitation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Professor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College, Huazhong, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided